CLINICAL TRIAL: NCT06614218
Title: Minimally Invasive Micro Sclerostomy (MIMS®) Retrospective Chart Review
Brief Title: MIMS® Retrospective Chart Review
Status: Not yet recruiting | Type: Observational
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MMS-EEU-9
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Open Angle Glaucoma
Keywords: Polypharmacy; Intraocular Pressure; MIMS; Minimally Invasive Glaucoma Surgery; MIGS; MTMT; Trabeculectomy; Sclerostomy
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIMS Surgery Cohort: This cohort consists subjects treated with MIMS® Device as a standalone procedure during time period (27 Sep 2023 - 31 May 2025), and with documented post-operative follow-up available in the medical charts.
  Interventions: Device: Minimally Invasive Micro Sclerostomy

INTERVENTIONS:
Device: Minimally Invasive Micro Sclerostomy — The MIMS® procedure uses the proprietary MIMS® device, which creates a sclerostomy in the eye.
  Other Names: MIMS

SUMMARY:
This is a post-market clinical follow-up, retrospective chart review of MIMS® surgical procedures conducted during time period between Sep 2023 and May 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Eye treated with MIMS® Device as a standalone procedure
2. MIMS® surgery was performed between 27 Sep 2023 and 30 April 2024

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects of Armenian descent that were treated with the MIMS® Device as a standalone procedure between 27 Sep 2023 and 30 April 2024.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in IOP from medicated baseline at 12 months post-MIMS® surgery | Medicated baseline at 12 months post-MIMS® surgery
Change in the number of topical IOP-lowering medications from medicated baseline at 12 months post-MIMS® surgery | Medicated baseline at 12 months post-MIMS® surgery
Success rate at 12 months post-MIMS® surgery | 12 months post-MIMS® surgery

CONTACTS AND LOCATIONS:
Locations (1):
- S. Malayan Eye Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided